CLINICAL TRIAL: NCT03054272
Title: Visual Perception Exploration Using Eye-tracking Technology in a Cannot Intubate/Cannot Oxygenate Simulation
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Issam Tanoubi, Université de Montreal, Université de Montréal
Other Study IDs: Expertise-2016
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Patient Simulation; Perception; Intubation; Difficult or Failed
Keywords: High-fidelity simulation; Eye-tracking; Difficult intubation
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents: Anesthesia residents from University of Montreal Anesthesia Department who were watching the video
  Interventions: Behavioral: Video
- Attending Physicians: Attending physicians from University of Montreal Anesthesia Department who were watching the video
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — A 13-minute video based on a suggested CICO algorithm from the Difficult Airway Society that was produced at the University of Montreal Simulation Centre using high-fidelity settings.

SUMMARY:
Using eye-tracking technology, the aim of this observational study is to compare the visual interests between attending physicians and residents watching a Cannot Intubate/Cannot Oxygenate (CICO) scripted and simulated scenario

DETAILED DESCRIPTION:
Attending physicians and residents, from the department of Anesthesiology at the Université de Montréal were recruited on a voluntary basis. A 13-minute video based on a suggested CICO algorithm from the Difficult Airway Society to manage unanticipated difficult intubation in adults (3) was produced at the University of Montreal Simulation Centre using high-fidelity settings. The scenario was about a patient, with a cervical collar, in the post-anesthesia care unit. Throughout the video, the patient presents increasing respiratory distress worsening to respiratory failure. The anesthesiologist fails to ventilate, intubate and insert a laryngeal mask leading to a cricothyroidotomy. All participants were looking at a screen on which the scenario was broadcast. The screen was equipped with TobiiEyeX®, an eye-tracking system that automatically aggregates gaze data.

ELIGIBILITY:
Inclusion Criteria:

* Residents and attending physicians from University of Montreal Anesthesia Department

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and attending physicians from University of Montreal Anesthesia Department
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Difference between Time to First Fixation and Total View Duration of areas of interests. | The primary endpoint is collected during 15 minutes, throughout the viewing of the video by the participant
  The screen was equipped with TobiiEyeX®, an eye-tracking system that automatically aggregates gaze data. The display was divided in seven Areas of Interest (AOI). Data were collected using the Tobii Studio® program to obtain the total view duration (TVD) of the various AOIs.

CONTACTS AND LOCATIONS:
Overall Officials: Issam Tanoubi, Dr, Study Director — Université de Montreal; Komi Sodoke, Msc, Principal Investigator — Université de Montreal; Mathieu Tourangeau, Dr, Principal Investigator — Université de Montreal

IPD SHARING:
Plan to Share IPD: No